CLINICAL TRIAL: NCT04388137
Title: Multi-center Study on the Establishment of Diagnostic Criteria System for Pediatric Functional Gastrointestinal Disorders in Mainland China
Brief Title: Multi-center Study on Pediatric Functional Gastrointestinal Disorders in Mainland China
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Mizu Jiang, Director of National Clinical Research Center for Child Health, Zhejiang University
Other Study IDs: MZJiang
Record Dates: First submitted 2020-04-19; First posted 2020-05-14 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: Functional Gastrointestinal Disorders
Keywords: functional gastrointestinal disorders; children
MeSH Terms: conditions — Gastrointestinal Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- infants aged 0-3: No intervention.
  Interventions: Other: No intervention.
- children aged 4-18: No intervention.
  Interventions: Other: No intervention.

INTERVENTIONS:
Other: No intervention. — No intervention.

SUMMARY:
This study plans to understand the prevalence and clinical characteristics of pediatric functional gastrointestinal disorders in mainland China through multi-center investigation and clinical epidemiological analysis, to reveal the prevalence characteristics and related factors of functional gastrointestinal disorders in children of all ages in mainland China, to establish a diagnostic standard system for pediatric functional gastrointestinal disorders in mainland China, to provide evidence-based basis for the formulation of new Roman standard for functional gastrointestinal disorders, and to provide new ideas and treatment basis for the diagnosis and treatment of functional gastrointestinal disorders in children.

DETAILED DESCRIPTION:
Functional gastrointestinal disorders (FGIDs), also known as brain-intestinal interaction abnormalities, are associated with dynamic disorders, high visceral sensitivity, changes in mucosal and immune functions, changes in intestinal flora, and abnormal central nervous system regulatory functions. FGIDs are the most common causes of diagnosis and treatment of gastrointestinal diseases in children. During the past 10 years, new progress has been made in the study of various FGIDs in children of different ages. FGIDs Rome Commission of Experts revised the relevant diagnostic criteria and officially published the Rome IV criteria for pediatric FGIDs in Gastroenterology in 2016. Due to many factors, the epidemiological survey data of pediatric FGID are still lacking in China. Whether Rome II, Rome III or Rome IV, their diagnostic criteria and epidemiological data were from other countries and regions, so their suitability for China's children remains to be verified. This study plans to understand the prevalence and clinical characteristics of pediatric functional gastrointestinal disorders in mainland China through multi-center investigation and clinical epidemiological analysis, to reveal the prevalence characteristics and related factors of functional gastrointestinal disorders in children of all ages in mainland China, to establish a diagnostic standard system for pediatric functional gastrointestinal disorders in mainland China, to provide evidence-based basis for the formulation of new Roman standard for functional gastrointestinal disorders, and to provide new ideas and treatment basis for the diagnosis and treatment of pediatric functional gastrointestinal disorders.

ELIGIBILITY:
Inclusion Criteria:

* Children diagnosed with functional gastrointestinal disorders

Exclusion Criteria:

* Children not diagnosed with functional gastrointestinal disorders

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children who visit the gastroenterology department due to gastrointestinal symptoms
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
the prevalence rate | From date of finishing the disease diagnosis until the date of statistical analysis completed, assessed up to 6 months
  the prevalence rate of pediatric functional gastrointestinal disorders in mainland China

SECONDARY OUTCOMES:
the Rome IV questionnaire | From date of finishing the questionnaire until the date of statistical information completed, assessed up to 3 months
  to understand the clinical characteristics of pediatric functional gastrointestinal disorders in mainland China

CONTACTS AND LOCATIONS:
Overall Officials: Mizu Mizu, Doctor, Principal Investigator — National Clinical Research Center for Child Health

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rouster AS, Karpinski AC, Silver D, Monagas J, Hyman PE. Functional Gastrointestinal Disorders Dominate Pediatric Gastroenterology Outpatient Practice. J Pediatr Gastroenterol Nutr. 2016 Jun;62(6):847-51. doi: 10.1097/MPG.0000000000001023. PMID 26513617
- [Background] Benninga MA, Faure C, Hyman PE, St James Roberts I, Schechter NL, Nurko S. Childhood Functional Gastrointestinal Disorders: Neonate/Toddler. Gastroenterology. 2016 Feb 15:S0016-5085(16)00182-7. doi: 10.1053/j.gastro.2016.02.016. Online ahead of print. PMID 27144631
- [Background] Robin SG, Keller C, Zwiener R, Hyman PE, Nurko S, Saps M, Di Lorenzo C, Shulman RJ, Hyams JS, Palsson O, van Tilburg MAL. Prevalence of Pediatric Functional Gastrointestinal Disorders Utilizing the Rome IV Criteria. J Pediatr. 2018 Apr;195:134-139. doi: 10.1016/j.jpeds.2017.12.012. Epub 2018 Feb 3. PMID 29398057
- [Background] Saps M, Moreno-Gomez JE, Ramirez-Hernandez CR, Rosen JM, Velasco-Benitez CA. A nationwide study on the prevalence of functional gastrointestinal disorders in school-children. Bol Med Hosp Infant Mex. 2017 Nov-Dec;74(6):407-412. doi: 10.1016/j.bmhimx.2017.05.005. Epub 2017 Sep 1. PMID 29382524